CLINICAL TRIAL: NCT01815593
Title: A Prospective, Randomized Study of Enhanced External Counterpulsation for Patients With Erectile Dysfunction
Brief Title: The Value of Enhanced External Counterpulsation on Erectile Dysfunction
Acronym: EECPED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chen Sheng Fu,MD, Principal Investigator, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EECPED
Record Dates: First submitted 2013-03-16; First posted 2013-03-21 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Vascular Endothelium; Counterpulsation, External
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: Patients with erectile dysfunction are assigned to two groups in parallel for the duration of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced External Counterpulsation (Experimental): Men with erectile dysfunction receive Enhanced External Counterpulsation treatment
  Interventions: Device: Enhanced external counterpulsation
- Control (No Intervention): Men with erectile dysfunction without Enhanced External Counterpulsation treatment

INTERVENTIONS:
Device: Enhanced external counterpulsation — Enhanced external counterpulsation therapy is done by sequential inflation of 3 sets of cuffs wrapped around the lower extremities during diastole and deflation of the cuffs during systole. The systolic deflation/ Diastolic inflation sequence of EECP leads to systolic unloading and diastolic augmentation, resulting in increased blood flow in a pulsatile manner. The patients receive 35-36 hours EECP intervention, 1 -hour session every day over a 7-week period.
  Other Names: EECP
  Arms: Enhanced External Counterpulsation

SUMMARY:
The purpose of this study is to investigate the efficacy of Enhanced External Counterpulsation (EECP) in patients with erectile dysfunction

DETAILED DESCRIPTION:
Patients with erectile dysfunction will be randomized into two groups: EECP intervention or not. Erectile function, hemodynamic parameters, vascular endothelial function will be measured and compared.

ELIGIBILITY:
Inclusion Criteria:

1. men over 18 years old;
2. provide signed informed consent;
3. existence of erectile dysfunction
4. agree not to use any other erectile dysfunction treatment at least one month;

Exclusion Criteria:

1. history of long drug abuse;
2. pelvic, spine, brain trauma or surgery;
3. endocrine, liver, lung, kidney disease, malignancies, hematological disorders;
4. abnormal urogenital status, such as small testicle (<2cm), penile plaques;

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-04 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Erectile function evaluated by International Index of Erectile Function-5 questionnaire | 7 weeks

SECONDARY OUTCOMES:
Endothelial function | 7 weeks
  Flow-mediated dilation：In this method,brachial artery diameter is measured before and after an increase in shear stress that is induced by reactive hyperemia (FMD). Endothelial progenitor cells：Flow cytometry to detect changes in the number of endothelial progenitor cells

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhang, M. D., Study Director — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Sakka A, Morsy A, Fagih B. Enhanced external counterpulsation in patients with coronary artery disease-associated erectile dysfunction. Part I: effects of risk factors. J Sex Med. 2007 May;4(3):771-779. doi: 10.1111/j.1743-6109.2007.00458.x. Epub 2007 Apr 13. PMID 17433083